CLINICAL TRIAL: NCT03165045
Title: AERIAL®: Changes in Health and Functional Status in Patients With COPD During Therapy With Spiolto® Respimat®
Brief Title: Changes in Health and Functional Status in Patients With Chronic Obstructive Pulmonary Disease During Therapy With Spiolto® Respimat® (AERIAL®)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0065
Record Dates: First submitted 2017-05-11; First posted 2017-05-24 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients treated with Spiolto® Respimat®: Patients with COPD
  Interventions: Drug: Spiolto® Respimat®

INTERVENTIONS:
Drug: Spiolto® Respimat® — 6 weeks
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO

SUMMARY:
The objective of this NIS is to measure changes in health status including functional status using CCQ scores in COPD patients receiving treatment with Spiolto® Respimat® according to label after approximately 6 weeks in routine clinical practice.

DETAILED DESCRIPTION:
The objective of this NIS is to measure changes in health status including functional status using CCQ scores in COPD patients receiving treatment with Spiolto® Respimat® according to label after approximately 6 weeks in routine clinical practice.

In visit 1, patient data on demographics, smoking status, medical history, breathlessness, general condition, health and functional status and adverse drug reactions will be collected. In visit 2, after approximately 6 weeks, data on smoking status, concomitant diseases and medication, general condition, health and functional status and adverse drug reactions will be collected; additionally data on patient satisfaction, continuation or discontinuation of treatment and the reason in case of discontinuation.

ELIGIBILITY:
Inclusion Criteria:

Patients can be included if all of the following criteria are met:

* Written informed consent prior to participation
* Female and male patients ≥40 years of age
* Patients diagnosed with COPD and requiring a combination of two long-acting bronchodilators (LAMA + LABA) according to approved SmPC and GOLD COPD guideline recommendation 2017 (GOLD COPD groups B to D)
* Treatment with Spiolto® Respimat® acc. to SmPC at the discretion of the physician.

Exclusion Criteria:

* Patients with contraindications according to Spiolto® Respimat® SmPC
* Patients already on a LABA/LAMA combination (free and fixed dose) in the last 6 weeks before study entry
* Patients continuing LABA-ICS treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
* Pregnancy and lactation
* Current participation in any clinical trial or any other non-interventional study of a drug or device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: approximately 1300 patients from approximately 400 sites in Germany will be collected. Site selection will be performed to reflect routine COPD care in Germany in order to secure representativeness of the COPD population.
Sampling Method: Probability Sample
Enrollment: 1351 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Marseille, 49613277141881, Study Chair — andrea.marseille@boehringer-ingelheim.com
Locations (108):
- Germany (108):
  - Dr. Weghmann, Aachen
  - Praxis Edgar Schaubert, Aldenhoven
  - MZM Medizin Zentr. Marienstrasse, Aldenhoven B Jülich
  - Praxis Dr. Selbig, Ansbach
  - Dr. Ludwig, Bad Bentheim
  - Dr. Jung, Bad Ditzenbach
  - Praxis Dr. med. Graubner, Bad Sachsa
  - Dr. Callitsis, Bad Vilbel
  - Dr. Junggeburth, Bad Wörishofen
  - Praxis Edgar Hossbach, Berkatal-Frankershausen
  - Dr. Urban, Berlin
  - Praxis Abdullah Sahan, Berlin
  - Dr. Kopf, Berlin
  - Dr. Thalhofer, Berlin
  - Gemeinschaftspraxis Dres. Wetterau/Dimar, Biberach
  - Dr. Kassik, Bitterfeld-Wolfen
  - Dr. Biedermann, Blankenhain , Thür
  - Praxis Dr. Andreas Schwittay, Böhlen
  - Gemeinschaftspraxis Dres. Bartels, Breuberg
  - Dres. Ottlewski/Sutor, Burgwedel
  - Praxis B. Metzlaff, Büchen
  - Praxis A. Hermann/L. Hermann, Cloppenburg
  - Praxis Dr. Käßner, Cottbus
  - Dres. Forster/Kneser/Steinmetz, Darmstadt
  - Dres. Jung/Jung, Deggingen
  - Dr. Franz, Dietzenbach
  - Dres. Tietjens/Tobias, Dortmund
  - Dr. Schwiese, Duisburg
  - Dr. Kontny, Duisburg
  - Dres. Berger/Schäfer/Winkels, Düren
  - Gemeinschaftspraxis Dres. Rommelmann/Lange/Geist/Neise, Düsseldorf
  - Ges. f. Med. Fortbildung, Düsseldorf
  - Praxis Dr. Andreas Kroll, Einbeck
  - Dr. Schmidt, Erfurt
  - Dres. Brüning/Schax, Essen
  - Praxis Dr. Schmorell, Forchheim
  - Dres. Engelhard/Wihl, Frankenberg
  - Studienzentrum Dr. Klaus Keller, Frankfurt
  - Dr. Morgner, Freiberg
  - Allgemeinmedizinische Gemeinschaftspraxis Dres. Fischer/Fischer, Friedrichsthal
  - Dr. Xanthopoulos, Fürstenwalde
  - Praxis A. Heinze, Fürstenwalde
  - Dr. Sommer, Garmisch-Partenkirchen
  - Praxis C. Staack/Z. Zadrozny, Gelsenkirchen
  - Praxis Dr. Körössy, Geretsried
  - Das HausarztZentrum, Grafenrheinfeld
  - Dres. Koenen & Partner, Grafenrheinfeld
  - Praxis Dr. med. Werner Gams, Gütersloh
  - Dr. Waida, Haan
  - Pneumologicum Halle, Halle
  - Praxis J. Lemke, Halle
  - Dr. Polke, Hamburg
  - Praxis Dr. Kaase, Hamburg
  - Dr. Abenhardt, Heidelberg
  - Praxis J. Hinrichs-Pavlik, Heidelberg , Neckar
  - Praxis Dr. Constance Koch, Heilbad Heiligenstadt
  - Praxis J. Korsakas, Heudeber
  - Praxis Dres. Berg & Partner, Höchstadt an der Aisch
  - Dr. Schulze, Jerichow
  - Ambulantes Zentrum, Kalawa
  - Dr. Schmitz, Kall
  - Praxis Dr. Bernhard Beckmann, Kamen
  - Praxis G. Mohanty, Kamp-Lintfort
  - Praxis Dr. Dietrich Auge, Koblenz
  - Dres. Lehmann/Schwerdtfeger, Köthen
  - Praxis Dr. Astrid Pfitzer, Kronach
  - KMG Klinikum Mitte GmbH, Kyritz , Prignitz
  - Praxis Dr. Weberling, Lahnau
  - POIS Leipzig GbR, Leipzig
  - Dres. Bonitz/Hoheisel, Leipzig
  - Dr. Seiz, Leonberg , Württ
  - Praxis Dr. Hannelore Pitule, Ludwigshafen am Rhein
  - Dres. Kock & Partner, Mainaschaff
  - Dr. Saur, Mannheim
  - Praxis Dr. Hermann A. Trauth, Marburg
  - Gemeinschaftspraxis Dres. Jansen/Nolzen, Menden
  - Dr. Bartsch, Moers
  - Dr. Schipper, Monheim
  - Praxis Hermann Ingerl, Mosbach
  - Praxis Dr. Jan Feimer, München
  - Thoraxzentrum Bez. Unterfranken, Münnerstadt
  - Praxis Dipl. med Thomas Hagen, Neumarkt
  - Praxis Wanda Wuttke, Nuremberg
  - Praxis Dr. Volker E. Trapp, Nuremberg
  - Praxis Dipl.-med. Anne-Kathrin Schmidt, Oschatz
  - Dr. Bauer, Potsdam
  - Praxis Dr. Rudolf Hennig, Radebeul
  - Dr. Jasch-Hoppe, Rathenow
  - Zentrum für Onkologie, Rostock
  - Dres. Herold/Kaa, Roth , Mittelfr
  - Lungenfachzentrum Rhein-Main, Rüsselsheim am Main
  - MVZ für Atemwegserkrankungen, Schleswig
  - Praxis S. Theuer, Seelow
  - Dres. Knöbel/Olesch/Pelz-Knöbel, Straubing
  - Dr. Eisenschmidt, Strausberg
  - Dr. Schröter, Trier
  - Dres. Barczok & Kollegen, Ulm, Donau
  - Dres. Günther/Günther, Viernheim
  - Überörtliche Gemeinschaftspraxis Dr. med. Albert Esselmann, Warendorf
  - Dres. Herold/Kaa, Weißenburg I Bay
  - Dres. Geissler/Geissler, Weißenfels, Saale
  - Dres. Seidel/Röcher, Wiefelstede
  - Dres. Fried/Thomas, Wiesbaden
  - Praxis K.P. Schaps/H. Zimmeck, Wilhelmshaven
  - Dr. Franz, Witten
  - Dr. Weber, Witten
  - Praxis D. Kubitscheck, Wittenberg
  - Dr. Riegel, Wolfsburg

REFERENCES:
- [Derived] Gillissen A, Marseille A, Skowasch D, Ritz J, Mattiucci-Guehlke M, Pabst S, Greulich T, Koczulla R. Health and functional status of tiotropium/olodaterol-treated patients with COPD: results from the AERIAL(R) non-interventional study. ERJ Open Res. 2021 Sep 6;7(3):00004-2021. doi: 10.1183/23120541.00004-2021. eCollection 2021 Jul. PMID 34513983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic obstructive pulmonary disease patients receiving treatment with Spiolto® Respimat® for approximately 6 weeks in routine clinical practice
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist site to ensure that they (the subjects) met all implemented inclusion/exclusion criteria.
Groups:
- Spiolto® Respimat®: Spiolto® Respimat® 2.5 microgram/2.5 microgram per puff inhalation solution Baseline visit at the start of the study
Period: Visit 1
Arm/Group | Spiolto® Respimat®
Started | 1351
Completed | 1322
Not Completed | 29
Not completed — No registration after visit 1 | 9
Not completed — No treatment documented | 10
Not completed — No visit 1 | 10
Period: Visit 2
Arm/Group | Spiolto® Respimat®
Started | 1322
Completed | 1140
Not Completed | 182
Not completed — Available CCQ score at visit 1 only | 109
Not completed — No available total CCQ score at all | 29
Not completed — Available total CCQ score at vist 2 only | 44

BASELINE CHARACTERISTICS:
Population: All patients who had given their written informed consent to study participation and at least one documented administration of Spiolto® Respimat® were included in the Treated Set (TS).
Groups:
- Spiolto® Respimat® at Study Start: Spiolto® Respimat® 2.5 microgram/2.5 microgram per puff inhalation solution Baseline visit at the start of the study
Arm/Group | Spiolto® Respimat® at Study Start
Number analyzed (Participants) | 1322
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.63 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 562
  Male | 760
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
CCQ Score [Mean (Standard Deviation); unit: Score] — Each of the 10 Clinical chronic obstructive pulmonary disease questionaire (CCQ) questions is scored by the patient on a 7-point scale between 0 (Never/Not limited at all) and 6 (Almost all the time/Totally limited or unable to do). The (total) CCQ score measures the health and functional status. Population: CCQ at baseline is measured for patients with an observation of the score for visit 1 and visit 2.
  Score
    Symptom (Items: 1; 2; 5; 6): number analyzed (Participants) | 1140
    Symptom (Items: 1; 2; 5; 6) | 3.42 (1.13)
    Functional state (CCQ-4) (Items: 7-10): number analyzed (Participants) | 1140
    Functional state (CCQ-4) (Items: 7-10) | 3.05 (1.24)
    Mental state (Items: 3; 4): number analyzed (Participants) | 1140
    Mental state (Items: 3; 4) | 2.69 (1.58)
    Total CCQ score (All subscales): number analyzed (Participants) | 1140
    Total CCQ score (All subscales) | 3.12 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Success
Description: The primary endpoint of the study was "therapeutic success" at visit 2.
  The CCQ questionnaire contained 10 questions about symptoms, functional status and mental status. Each of the 10 CCQ questions was scored by the patient on a 7-point scale between 0 and 6 at baseline and at the end of observation after approximately 6 weeks. The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. A higher CCQ score is indicative of worse status. A decrease of 0.4 points is considered to be the minimal clinically important difference (MCID) for both CCQ score and CCQ-4.
Time Frame: Final visit at the end of the study, approximately 6 weeks after start of study
Population: All screened patients with informed consent, at least one documented administration of Spiolto® Respimat® and available CCQ scores at visit 1 and visit 2, were defined as full analysis set (FAS).
Measure: Count of Participants; unit: Participants
Groups:
- Spiolto® Respimat: Spiolto® Respimat® 2.5 microgram/2.5 microgram per puff inhalation solution
Arm/Group | Spiolto® Respimat
Number analyzed (Participants) | 1140
Participants
  Therapy successfull | 756

2. Secondary Outcome: Assessment of Changes in CCQ and CCQ-4 From Visit 1 to Visit 2
Description: Absolute changes in total CCQ score and CCQ-4 score from baseline visit at the start of the study to final visit at the end of study.
  The CCQ questionnaire contained 10 questions about symptoms, functional status and mental status. The sum of the scores divided by 10 gives the CCQ score which measures the health and functional status. A higher CCQ score is indicative of worse status. A change of 0.4 points is was considered to be the minimal clinically important difference (MCID) for both CCQ score and CCQ-4.
Time Frame: Final visit at the end of the study, approximately 6 weeks after start of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of patients (%)
Arm/Group | Spiolto® Respimat
Number analyzed (Participants) | 1140
Percentage of patients (%)
  Symptom | 0.84 (1.06)
  Functional State (CCQ-4) | 0.75 (1.05)
  Mental state | 0.73 (1.34)
  Total CCQ Score | 0.78 (0.95)

3. Secondary Outcome: General Condition of the Patient
Description: General condition of the patient, evaluated by the physician (Physician's global Evaluation score) at visit 1 and visit 2.
  The treating physician used the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent). The modified Medical Research Council (mMRC) scale was used to assess the breathlessness state of the patient before the treatment.
Time Frame: Baseline visit (Visit 1) at the start of the study and final visit at the end of the study (visit 2), approximately 6 weeks after visit 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Spiolto® Respimat® Final Vist: Spiolto® Respimat® 2.5 microgram/2.5 microgram per puff inhalation solution
Arm/Group | Spiolto® Respimat® at Study Start | Spiolto® Respimat® Final Vist
Number analyzed (Participants) | 1140 | 1140
Participants
  Score 1 | 11 | 1
  Score 2 | 93 | 23
  Score 3 | 281 | 95
  Score 4 | 378 | 223
  Score 5 | 195 | 350
  Score 6 | 138 | 325
  Score 7 | 43 | 102
  Score 8 | 1 | 20
  Missing | 0 | 1

4. Secondary Outcome: Patient Satisfaction With Spiolto® Respimat® at Visit 2
Description: A patient satisfaction survey was performed at visit 2, using a 7-point ordinal scale with divisions from very dissatisfied to very satisfied.
  The 7-item satisfaction scale is a self-designed Boehringer-Ingelheim scale, without a public source or validation status.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat
Number analyzed (Participants) | 1140
Participants
  Patient overall satisfaction: Very satisfied | 427
  Patient overall satisfaction: Satisfied | 544
  Patient overall satisfaction: Rather satisfied | 95
  Patient overall satisfaction: Neither satisfied nor dissatisfied | 46
  Patient overall satisfaction: Rather dissatisfied | 13
  Patient overall satisfaction: Dissatisfied | 12
  Patient overall satisfaction: Very dissatisfied | 3
  Patient satisfaction with inhaling: Very satisfied | 429
  Patient satisfaction with inhaling: Satisfied | 579
  Patient satisfaction with inhaling: Rather satisfied | 85
  Patient satisfaction with inhaling: Neither satisfied nor dissatisfied | 33
  Patient satisfaction with inhaling: Rather dissatisfied | 8
  Patient satisfaction with inhaling: Dissatisfied | 4
  Patient satisfaction with inhaling: Very dissatisfied | 2
  Patient satisfaction with handling: Very satisfied | 389
  Patient satisfaction with handling: Satisfied | 590
  Patient satisfaction with handling: Rather satisfied | 116
  Patient satisfaction with handling: Neither satisfied nor dissatisfied | 24
  Patient satisfaction with handling: Rather dissatisfied | 16
  Patient satisfaction with handling: Dissatisfied | 4
  Patient satisfaction with handling: Very dissatisfied | 1

5. Secondary Outcome: Number of Participants Willing to Continue Treatment With Spiolto® Respimat® at Visit 2
Description: To assess the willingness to continue treatment with Spiolto® Respimat® at visit 2 patients were asked a yes/no question if they would continue the treatment.
Time Frame: 6 weeks
Population: Patients with a performed visit 2
Measure: Count of Participants; unit: Participants
Arm/Group | Spiolto® Respimat
Number analyzed (Participants) | 1254
Participants | 1194

ADVERSE EVENTS:
Time Frame: approximated up to 6 weeks after visit 1
Groups:
- Total: Spiolto® Respimat® 2.5 microgram/2.5 microgram per puff inhalation solution
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 1/1322
Serious Adverse Events (participants affected / at risk) | 1/1322
Other Adverse Events (participants affected / at risk) | 0/1322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=1322)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03165045/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT03165045/SAP_001.pdf